CLINICAL TRIAL: NCT01833208
Title: Pilot: Impact of High-Dose, Single Fraction Radiation on Immunogenicity of Sipuleucel-T in Metastatic Castration Recurrent Prostate Cancer Patients
Brief Title: Radiation Therapy in Treating Patients With Metastatic Hormone-Resistant Prostate Cancer Receiving Sipuleucel-T
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: Dendreon (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I 223912; NCI-2013-00633 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 223912 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2013-04-02; First posted 2013-04-16 (Estimated); Last update posted 2021-08-05 (Actual); Status verified 2021-08

CONDITIONS: Hormone-Resistant Prostate Cancer; Metastatic Malignant Neoplasm in the Bone; Recurrent Prostate Carcinoma; Stage IV Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment (radiation therapy) (Experimental): Patients undergo single-fraction radiation therapy to at least 1 bone lesion 2 days after the first sipuleucel-T dose.
  Interventions: Other: Laboratory Biomarker Analysis; Radiation: Radiation Therapy

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Radiation: Radiation Therapy — Undergo single-fraction radiation therapy
  Other Names: Cancer Radiotherapy; Irradiate; Irradiated; Irradiation; RADIATION; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation

SUMMARY:
This pilot clinical trial studies the impact of radiation therapy on the immunogenicity of Sipuleucel-T. Patients with castration recurrent prostate cancer who are eligible for treatment with Sipuleucel-T and who have bone metastases are eligible.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess whether radiation therapy (RT) increases the immunogenic potential or sipuleucel-T in participants with castration recurrent prostate cancer.

II. To assess systemic changes to the immune system and genetic changes to immune cells in participants treated by the combination of RT and sipuleucel-T.

III. To assess the induction of antigen-specific immune responses to prostatic acid phosphatase (PAP), cancer/testis antigen 1B (NY-ESO-1) and antigens that have proven to be released by radiation (such as, heat shock protein 90 [HSP-90], calreticulin, etc.).

SECONDARY OBJECTIVES:

I. To assess adverse event rates in participants receiving the high-dose radiation and sipuleucel-T therapy.

II. To assess prostate-specific antigen (PSA) changes. III. To assess overall and cancer specific survival.

OUTLINE:

Patients undergo single-fraction radiation therapy to at least 1 bone lesion 2 days after the first sipuleucel-T dose.

After completion of study treatment, patients are followed up at 3 and 6 months and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Have minimally symptomatic metastatic castration recurrent prostate cancer with bone lesions; this patient population is defined as having failed hormone treatment and has insurance approval for PROVENGE® therapy
* Patients that have been prescribed sipuleucel-T and have not started treatment
* Must be candidates for radiation treatment to bone lesions
* Patient or legal representative must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of =< 2

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study
* Patients who have received prior radiation of osseous lesions
* Patients who have received any prior immunotherapy
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Unwilling or unable to follow protocol requirements
* Any condition which in the investigator's opinion deems the patient an unsuitable candidate

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2013-07-03 (Actual); Primary Completion 2018-08-06 (Actual); Study Completion 2021-01-23 (Actual)

PRIMARY OUTCOMES:
Capacity of T cells to proliferate in response to antigen stimulation, assessed with a tritiated thymidine incorporation assay and an interferon-gamma enzyme-linked immunosorbent spot assay | Up to 6 months
  Will be assessed using Wilcoxon Signed Rank and McNemar's tests for continuous and dichotomous endpoints respectively.
Change in antigen-specific humoral response measured via enzyme-linked immunosorbent assay | Baseline up to 6 months
  Will be assessed using Wilcoxon Signed Rank and McNemar's tests for continuous and dichotomous endpoints respectively.
Change in the genetics of immune effectors, measured with ribonucleic acid from monocytic and lymphocytic cells | Baseline to 6 months
  Will be assessed using Wilcoxon Signed Rank and McNemar's tests for continuous and dichotomous endpoints respectively.
Quantification of lymphocyte subsets and NK cells | Baseline to 6 months
  Will be assessed using Wilcoxon Signed Rank and McNemar's tests for continuous and dichotomous endpoints respectively.

SECONDARY OUTCOMES:
Adverse event rates assessed using National Cancer Institute Common Terminology Criteria for Adverse Events version 4 | Up to 6 months
  The Clopper-Pearson one-sided upper 95% confidence limit will be provided. Associations between baseline characteristics and presence of an adverse event will be considered using the Wilcoxon rank sum test (or Cochran-Armitage test for trend) and Fisher's exact test respectively. Bar charts, scatterplots and other descriptive and graphical methods will also be utilized.
Cancer-specific survival | Up to 2 years
  Will be depicted using Kaplan Meier methods.
Change in PSA | Baseline up to 6 months
Overall survival | Up to 2 years
  Will be depicted using Kaplan Meier methods.

CONTACTS AND LOCATIONS:
Overall Officials: Gurkamal Chatta, MD, Principal Investigator — Roswell Park Cancer Institute
Locations (2):
- United States (2):
  - Roswell Park Cancer Institute, Buffalo, New York
  - Western New York Urology Associates LLC-Harlem, Cheektowaga, New York